CLINICAL TRIAL: NCT06473506
Title: Exploring the Use of Saliva for the Detection of Group A Streptococcus
Brief Title: Group A Streptococcus Saliva Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Aaron Campigotto, Division Head Microbiology, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000081444
Record Dates: First submitted 2024-06-17; First posted 2024-06-25 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Group A Streptococcal Infections
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Saliva collection (Other): Self-collected saliva sample
  Interventions: Diagnostic Test: Saliva collection

INTERVENTIONS:
Diagnostic Test: Saliva collection — Self-collected saliva sample with molecular testing performed. Results are compared to rapid antigen testing, bacterial throat culture and bacterial throat molecular testing

SUMMARY:
This study is being done to evaluate whether saliva can be used to diagnose GAS infection and also to compare different testing methods in the microbiology lab. The saliva sample testing will be compared to the throat swab testing to see if saliva testing works as well. The lab will also try different testing methods to see if a faster type of testing (e.g. molecular testing) works as well as the regular method, which takes 48 hours to get results.

This is important because throat swabs can be challenging to collect in some children, and saliva is often much easier and more acceptable by children to collect. This could improve our ability to accurately diagnose and treat GAS infections.

ELIGIBILITY:
Inclusion Criteria:

* < 19 years of age
* Have provided a sample for GAS testing (bacterial throat swab or POCT rapid antigen test) at the discretion of the clinical team
* Able to provide a saliva sample

Exclusion Criteria:

* Parent/guardian and/or patient unable to consent or assent
* Unable to provide a saliva sample

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate and sensitivity of GAS detection | Within 24 hours of collection
  compare the rate and sensitivity of GAS detection by throat bacterial culture, throat molecular detection and saliva molecular detection according to a semi-quantitative value (quantified growth on bacterial culture or CT value for molecular assays)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Monica Caldeira-Kulbakas, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No